CLINICAL TRIAL: NCT00119470
Title: EUS-FNA in the Pre-Operative Evaluation of Patients With Lung Cancer: A Randomized Trial
Brief Title: EUS-FNA in the Pre-Operative Evaluation of Patients With Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004/276
Record Dates: First submitted 2005-07-01; First posted 2005-07-13 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: EUS-FNA
Procedure: Conventional Surgical Technique

SUMMARY:
This trial examines the role of EUS-FNA (Oesophageal Endoscopic Ultrasound with Fine Needle Aspiration) as an endoscopic technique for the mediastinal staging of patients with lung cancer.

Patients will be randomized to either conventional surgical technique or EUS-FNA.

ELIGIBILITY:
Inclusion Criteria:

* patients with histological or cytological proof of non small cell lung cancer (NSCLC) or with a high clinical suspicion for lung cancer (but without pathologically confirmed diagnosis from the bronchoscopy or CT guided transthoracal biopsies) in whom the next step is normally a diagnostic or therapeutic surgical intervention
* no distant metastases after routine clinical work up (PET is optional, not mandatory)
* provision of a written informed consent
* recent CT-scan of the thorax (<28 days before randomization date)
* age 18 years or older
* clinically fit for surgery

Exclusion Criteria:

* proof of small cell lung cancer (SCLC) with CWU (bronchoscopy or CT guided transthoracal punction)
* stage IV NSCLC
* patients with a solitary pulmonary nodule (thus without enlarged mediastinal lymph nodes on CT and without mediastinal PET hot spots) : these do not require further mediastinal investigation
* former therapy (chemotherapy or radiotherapy or surgery) for lung cancer
* other concomitant malignancies
* reasons for which the patient is unable to swallow the EUS-instrument (e.g. zenker diverticulum, unexplained esophageal stenosis)
* uncorrected coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Percentage of surgical interventions avoided

SECONDARY OUTCOMES:
Accuracy of EUS-FNA for mediastinal staging of lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Tournoy, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Tournoy KG, De Ryck F, Vanwalleghem LR, Vermassen F, Praet M, Aerts JG, Van Maele G, van Meerbeeck JP. Endoscopic ultrasound reduces surgical mediastinal staging in lung cancer: a randomized trial. Am J Respir Crit Care Med. 2008 Mar 1;177(5):531-5. doi: 10.1164/rccm.200708-1241OC. Epub 2007 Oct 25. PMID 17962631
- See also: Website University Hospital Ghent — http://www.uzgent.be